CLINICAL TRIAL: NCT03102970
Title: Morpho-COPD1b : Pain Assessment in Patients With Chronic Obstructive Pulmonary Disease (COPD) Exacerbations.
Brief Title: Pain Assessment in Patients With Chronic Obstructive Pulmonary Disease (COPD) Exacerbations.
Acronym: MorphoCOPD1b
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC15.324; DR-2016-269 (Other: CNIL)
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, Pain, Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of chronic obstructive pulmonary disease (COPD) is between 8 and 12% of the adult population. This prevalence is expected to increase over the coming decades due to the aging of the population and the continued exposure to risk factors for the disease. The evolution of COPD is marked by the occurrence of exacerbations of varying severity and patients are frequently admitted to the emergency department for evaluation, treatment and / or hospitalization. Admission in emergency department for COPD exacerbation represents approximately 1% of emergency admission.

Chronic pain is common in patients with Chronic Obstructive Pulmonary Disease (COPD). The pain intensity may increase during acute episodes of exacerbations. This study is aimed to compare pain intensity during exacerbation and stable phase of patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Chronic pain is common in patients with Chronic Obstructive pulmonary Disease (COPD). The pain intensity may increase during acute episodes of exacerbation. Fifty (50) patients in acute exacerbation of COPD will be included in the emergency department of CHU Grenoble Alpes and Hôpital du Sacré Coeur de Montréal. The intensity and characteristics of pain will be evaluated from the Short-Form McGill Pain Questionnaire (SF-MPQ) and the Brief Pain Inventory (BPI). Assessment of respiratory status, anxiety and depression, and clinical and biological data, defining the severity of exacerbation, will also be collected. A 30-day follow-up visit, after a return to the stable state of COPD, allowed the realization of Respiratory Functional Exploration and the same questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 years
* smoking at least ≥ 10 pack years
* previous FEV / FVC <0.70 post bronchodilator
* admitted for exacerbations (GOLD definition)

Exclusion Criteria:

* A dementia or non-communicating patient
* Patient with chronic pain of neoplastic origin or severe trauma (fracture , dislocation or severe pain) within 15 days before the date of inclusion
* Patient with no social security insurance , with restricted liberty or under legal protection
* Pregnant woman parturient or nursing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to emergency department for acute episodes of exacerbation of chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Variation of the short-form McGill Pain Questionnaire (SF-MPQ) between the exacerbation and the stable phase at 30 days | 30 days after exacerbation
  McGill Pain Questionnaire (SF-MPQ)

CONTACTS AND LOCATIONS:
Overall Officials: Maxime MAIGNAN, Principal Investigator — University Hospital, Grenoble
Locations (2):
- Emergency department of Hôpital du Sacré Coeur de Montréal, Montreal, Canada
- Emergency Department of university hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No